CLINICAL TRIAL: NCT03766490
Title: A Prospective, Single-arm, Multicenter Study of Anlotinib Hydrochloride Combined With First-generation EGFR TKIs as Second-line Treatment in Acquired (Non-T790M Mutation) Resistance Advanced Non-small Cell Lung Cancer
Brief Title: Anlotinib Hydrochloride Combined With EGFR TKIs in Advanced Non-small Cell Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: The First People's Hospital of Changzhou (Other); Second Affiliated Hospital of Soochow University (Other); Nantong University (Other); Affiliated Hospital of Jiangnan University (Other); Jiangyin People's Hospital (Other); Changzhou No.2 People's Hospital (Other); Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTER-L010
Record Dates: First submitted 2018-12-02; First posted 2018-12-06 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2018-12

CONDITIONS: Non-Small-Cell Lung
MeSH Terms: interventions — Gefitinib; icotinib

STUDY DESIGN:
Intervention Model Description: Anlotinib Hydrochloride Combined With gefitinib or Icotinib
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib Hydrochloride plus gefitinib or icotinib (Experimental)
  Interventions: Drug: Anlotinib Hydrochloride; Drug: Gefitinib; Drug: Icotinib

INTERVENTIONS:
Drug: Anlotinib Hydrochloride — Capsule, P.O. 12mg qd ,days 1-14, 21 days a cycle
Drug: Gefitinib — Tablet, P.O. 250mg qd
Drug: Icotinib — Tablet, P.O. 125mg tid

SUMMARY:
After the second-line treatment of patients with non-T790M mutations, chemotherapy with platinum-containing drugs was used, and chemotherapy-related toxicity was high. Studies have shown that bevacizumab combined with EGFR TKI have a good trend of benefit. This study is aimed to evaluate the efficacy and safety of Anlotinib Hydrochloride combined with first-generation EGFR TKIs as second-line treatment in advanced non-small cell lung cancer . The patients with IV non-small lung cancer have acquired resistance to prior first-generation EGFR TKIs and have non-T790M mutation.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histlogically confirmed stage IV non-small cell lung cancer .
* The initial treatment with gefitinib/icotinib evaluated PR/NC and the efficacy lasted for more than 6 months, then the disease progressed later. (The efficacy was assessed as PD according to the evaluation standard of RECIST1.1)
* At least a measurable lesion that meets the RECIST 1.1 criteria.
* Any gender. Age ≥18 years and ≤75 years
* Life expectancy >3 months.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1.
* Previously, EGFR gene test showed EGFR exon 19 deletion or exon 21 (L858R) mutation, and the gene test showed no T790M mutation before enrollment.
* Adequate organ function: haemoglobin ≥ 90 g/L;neutrophils count ≥1.5×109/L; platelet count ≥ 90 × 109/L; total bilirubin ≤ 1.5 × ULN ;ALT < 2 × ULN, (ALT < 5 × ULN, for those with liver metastases);AST < 2 × ULN, (AST < 5 × ULN, for those with liver metastases); Cr≤1.5× ULN.
* Echocardiography : LVEF≥50%
* 12-leads electrocardiogram : QTcF<450ms (man), <470ms(woman)
* Patient informed consent and signed written consent
* Patient compliance was good and voluntary follow-up, treatment, laboratory testing, and other research steps were performed as planned.

Exclusion Criteria:

* The patient has previously received anti-tumor therapy for EGFR TKIs other than gefitinib and ectinib for lung cancer.
* Patients that cannot detect EGFR gene, or patients with known T790M mutation.
* Small cell lung cancer (including lung cancer mixed with small cell lung cancer and non-small cell lung cancer).
* CT or MRI shows that the tumor lesion is ≤ 5 mm from the large vessel, or there is a central tumor that invades the local large blood vessel; or there is a significant pulmonary cavity or necrotizing tumor.
* Active brain metastasis, cancerous meningitis, spinal cord compression patients.
* Other active malignancies that require simultaneous treatment.
* Has a history of malignant tumors in the past 5 years.
* Patients with previous anti-tumor treatment-related adverse reactions who have not recovered to NCI-CTC AE≤1.
* Abnormal coagulation ,with bleeding tendency or undergoing thrombolysis or anticoagulant therapy.
* Renal insufficiency: urinary protein ≥ ++, or confirmed 24-hour urine protein ≥ 1.0g, or creatinine clearance <60ml / min.
* Severe acute or chronic infection requiring systemic treatment.
* Suffering from severe cardiovascular disease: myocardial ischemia ,myocardial or arrhythmia.
* Clinically significant hemoptysis occurred within 3 months prior to enrollment; or significant clinically significant bleeding symptoms or a clear tendency to hemorrhage.
* Untreated active hepatitis : Hepatitis B or Hepatitis C

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2019-03-30 (Estimated); Primary Completion 2019-12-20 (Estimated); Study Completion 2020-12-20 (Estimated)

PRIMARY OUTCOMES:
PFS（Progress free survival） | each 42 days up to PD or death(up to 24 months)
  PFS defined as the time from first dose of study treatment until the first date of either objective disease progression or death due to any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | From randomization until death (up to 24 months)
  OS is defined as the time until death due to any cause.
Objective Response Rate (ORR) | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  ORR is defined as the percentage of subjects with evidence of a confirmed complete response (CR) or partial response (PR) as per Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1.prior to progression or any further therapy.
Quality of Life(QoL) | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  use EORTC QLQ-C30(version 3) questionnaire to evaluate the quality of life.
Disease Control Rate (DCR) | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  Defined as the proportion of patients with a documented complete response, partial response, and stable disease (CR + PR + SD) based on RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Min Tao, Doctor, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated hospital of soochow university, Suzhou, Jangsu, China